CLINICAL TRIAL: NCT00429962
Title: Randomized, Phase IIIb Study Comparing Safety, Tolerability and Efficacy Between Lucentis® Administered in Conjunction With PDT With Visudyne® and Lucentis® in Patients With Subfoveal CNV Secondary to Age-Related Macular Degeneration
Brief Title: Study Comparing Ranibizumab Monotherapy With Combined Verteporfin Therapy in Subfoveal CNV
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Selim Orgul, University Hospital, Basel, Switzerland
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 081-PRC-2006-005
Record Dates: First submitted 2007-01-31; First posted 2007-02-01 (Estimated); Last update posted 2009-04-07 (Estimated); Status verified 2009-04

CONDITIONS: Choroidal Neovascularization; Age-Related Macular Degeneration
Keywords: subfoveal choroidal neovascularization (CNV); age-related macular degeneration; ranibizumab monotherapy; combined verteporfin-therapy; Lucentis® (ranibizumab); Visudyne®; photodynamic therapy
MeSH Terms: conditions — Choroidal Neovascularization; Macular Degeneration | interventions — Ranibizumab; Photochemotherapy; Verteporfin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): intravitreal ranibizumab used in combination with verteporfin photodynamic therapy
  Interventions: Drug: intravitreal ranibizumab & photodynamic therapy
- B (Active Comparator): intravitreal ranibizumab
  Interventions: Drug: intravitreal ranibizumab

INTERVENTIONS:
Drug: intravitreal ranibizumab — intraocular injection
  Other Names: Lucentis
  Arms: B
Drug: intravitreal ranibizumab & photodynamic therapy — intraocular injection photodynamic treatment (LASER) after intravenous injection
  Other Names: Visudyne
  Arms: A

SUMMARY:
This pilot study is designed to evaluate the safety and efficacy of intravitreal ranibizumab used in combination with verteporfin photodynamic therapy (Visudyne®) compared to ranibizumab monotherapy for the treatment of subfoveal CNV secondary to AMD

DETAILED DESCRIPTION:
Intravitreal ranibizumab has shown to increase average vision in patients with subfoveal CNV secondary to AMD. However, the treatment does not provide benefit to all patients and the treatment regimen requires monthly intravitreal injections. Ranibizumab is an anti-VEGF-A monoclonal antibody fragment. Verteporfin photodynamic therapy acts through occluding newly formed vessels. The combination of these therapies acting through different modes of action bears the potential to provide a more convenient and less frequent therapy while maintaining/improving the increase in vision improvement observed with ranibizumab monotherapy. The strategic goal is to evaluate whether intravitreal ranibizumab in combination with verteporfin photodynamic therapy is an effective, safe and convenient treatment for patients with subfoveal CNV secondary to AMD and explore potential advantages of such treatment compared to ranibizumab monotherapy

ELIGIBILITY:
Inclusion Criteria:

1. patients over 50 years, subfoveal CNV of any type secondary to age-related macular degeneration (AMD), no "macula-treatment for the last 30 days (e.g. with PDT, TA, Laser, Macugen®).

   * the area of the CNV must occupy at least >50% of the lesion (total lesion size under 5400 microns in greatest linear dimension)
   * Occult CNV:

     * recent disease progression
     * bleeding
     * VA decreased the last three months >5 letters or 2 or more than two lines (Snellen)
     * 10% increase of the lesion size the last three months
2. Best corrected visual acuity score between 24-73 letters (20/40 to 20/320) (ETDRS 4 m)

Exclusion Criteria:

1. Prior treatment with mit Laser, PDT, Macugen, TA
2. Prior treatment with radiatio, vitrectomy, transpupillary thermotherapy
3. History of surgical intervention in the study eye within two months preceding day 1
4. concurrent use of systemic anti-VEGF agents
5. previous treatment with or participation in a clinical trial involving anti-angiogenic drugs (Pegaptanib, ranibizumab, anecortave acetate of corticosteroids).
6. Ocular disorders in the study eye that may confound interpretation of the study results, including retinal detachment or macular hole (Stage 3 or 4), active intraocular inflammation (grade trace or above) or persistent macular edema due to uveitis or other inflammatory diseases
7. Retinal pigment epithelium tear, vitreous hemorrhage or history of rhegmatogenous retinal detachment or macular hole in the study eye
8. History of idiopathic or autoimmune-associated uveitis in either eye, active infectious conjunctivitis, keratitis, scleritis or endophthalmitis in either eye
9. Extracapsular extraction of cataract with phacoemulsification within two months preceding day 1, or a history of post-operative complications within the last 12 months preceding day 1 or a history of post-operative complications within the last 12 months preceding day 1 in the study eye (uveitis, cyclitis, iritis etc.)
10. Glaucoma with IOP>25 mmHg despite therapy
11. Aphakia or absence of the posterior capsule in the study eye
12. Spherical equivalent >-8

Ages: 50 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2006-07; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
First injection with PDT | monthly

SECONDARY OUTCOMES:
Monthly clinical evaluation of safety and necessity of re-intravitreal injection of ranibizumab after three initial injections | monthly

CONTACTS AND LOCATIONS:
Overall Officials: Ulrike Schneider, MD, Study Director — University Eye Clinic Basel
Locations (1):
- University Eye Clinic, Basel, Canton of Basel-City, Switzerland